CLINICAL TRIAL: NCT02227238
Title: A Phase 3b, Randomized, Open-label Study of the Antiviral Activity and Safety of Dolutegravir Compared to Lopinavir/Ritonavir Both Administered With Dual Nucleoside Reverse Transcriptase Inhibitor Therapy in HIV-1 Infected Adult Subjects With Treatment Failure on First Line Therapy
Brief Title: Comparative Efficacy and Safety Study of Dolutegravir and Lopinavir/Ritonavir in Second-line Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200304; 2014-001057-17 (EudraCT Number)
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
Keywords: integrase inhibitor; non-inferiority; dolutegravir; lopinavir/ritonavir; second-line treatment; HIV-1; antiretroviral therapy-experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DTG arm (Experimental): Subjects will receive one oral tablet of 50 mg DTG once daily plus two NRTIs selected by the investigator
  Interventions: Drug: DTG; Drug: Two NRTIs
- LPV/RTV arm (Active Comparator): Subjects will receive four oral tablets of200/50 mg LPV/RTV once daily or two oral tablets of 200/50 mg LPV/RTV twice daily plus two NRTIs selected by the investigator
  Interventions: Drug: LPV/RTV; Drug: Two NRTIs

INTERVENTIONS:
Drug: DTG — DTG is supplied as 50 mg tablets
  Arms: DTG arm
Drug: LPV/RTV — LPV/RTV is supplied as the LPV/RTV oral tablet, which contains 200 mg of LPV and 50 mg of RTV
  Arms: LPV/RTV arm
Drug: Two NRTIs — Investigators will choose a dual NRTI background regimen for each subject . In consultation with the medical monitor, 3TC may be added as a third NRTI to a dual-NRTI background regimen in subjects with chronic HBV infection and evidence of HIV resistance to 3TC

SUMMARY:
For treatment of human immunodeficiency virus type 1(HIV-1), publicly funded programmes tend to follow World Health Organization (WHO) guidelines to use a non-nucleoside reverse transcriptase inhibitor (NNRTI) combined with two nucleoside reverse transcriptase inhibitors (NRTIs) for first-line antiretroviral therapy (ART); however, there is a need for further data on the best treatment options for people with HIV-1 who have virological failure with this first-line regimen. The number of patients failing on their first-line regimen is increasing thereby requiring a switch to second-line treatment to reduce accumulation of drug-resistance mutations, disease progression, HIV transmission, and death. WHO guidelines recommend second-line antiretroviral therapy for adults consisting of two NRTIs + a ritonavir-boosted protease inhibitor (PI); atazanavir (ATV) plus ritonavir (RTV) or lopinavir (LPV)/RTV are the preferred boosted PI options. This study is conducted to demonstrate non-inferior antiviral activity at 48 weeks of a dolutegravir (DTG) containing regimen compared to a WHO-recommended standard of care regimen for second line treatment, LPV/RTV + two NRTIs, in HIV-1 infected patients failing first line therapy. This study comprises of a Screening Phase (approximately 28 to 42 days), a Randomized Phase (Day 1 to Week 48 plus a 4-week treatment extension), and a Continuation Phase. Approximately 612 subjects will be randomized 1:1 to receive DTG 50 milligram (mg) once daily or LPV/RTV (800/200 mg once daily or 400/100 mg twice daily, in accordance with investigator decision and local label), each added to an investigator selected background regimen of two NRTIs at least one of which needs to be fully active based on viral resistance testing at Screening. Subjects randomized to the LPV/RTV arm will either (i) continue receiving LPV/RTV and complete the study after the 4-week treatment extension at Week 52, or (ii) switch to the DTG arm prior to study completion at Week 52 and continue to have access to DTG in the Continuation Phase. Subjects randomized to receive DTG who successfully complete 52 weeks of treatment and subjects originally randomized to receive LPV/RTV but switched to DTG prior to Week 52 will continue to have access to DTG until it is either locally approved and commercial supplies are available to patients or the patient no longer derives clinical benefit, or the patient meets a protocol-defined reason for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected subjects >=18 years of age.
* A female subject may be eligible to enter and participate in the study if she:

is of non-childbearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and >=45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy, or bilateral oophorectomy or, is of child-bearing potential, with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the protocol-defined methods of contraception to avoid pregnancy throughout the study and for at least 2 weeks after discontinuation of all study medication.

* HIV-1 infection as documented by HIV-1 RNA >=400 c/mL at Screening.
* Subject has been on a first-line treatment regimen consisting of an NNRTI plus two NRTIs for at least 6 months and is currently experiencing virologic failure to this first-line regimen defined as two consecutive (>=7 days apart) HIV-1 RNA results of >=400 c/mL.
* Subjects must receive at least one fully active agent within the dual-NRTI background regimen for second line treatment. Fully active is defined by the Screening genotypic resistance report of the central laboratory (or a laboratory contracted by the central laboratory) showing no evidence of full or of partial resistance for a given NRTI which will be taken on study.
* Subject is PI-naïve and Integrase inhibitor (INI)-naïve, defined as no prior or current exposure to any PI or INI.
* Subject or the subject's legal representative is willing and able to understand and provide signed and dated written informed consent prior to screening.

Exclusion Criteria:

* Women who are breastfeeding.
* Any evidence of an active Centers for Disease Control and Prevention (CDC) Category C disease Exceptions include cutaneous Kaposi's sarcoma not requiring systemic therapy and historic or current CD4+ cell levels <200 cells per cubic millimeter
* Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Anticipated need for hepatitis C virus (HCV) therapy during the Randomized Phase of the study.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the subject.
* Subjects who in the investigator's judgment, poses a significant suicidality risk. Recent history of suicidal behavior and/or suicidal ideation may be considered as evidence of serious suicide risk.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Treatment with any of the following agents within 28 days of Screening: radiation therapy, cytotoxic chemotherapeutic agents, systemically administered immunomodulators.
* Treatment with any agent, other than licensed ART as allowed above with documented activity against HIV-1 in vitro/vivo within 28 days of first dose of IP. The exception is use of entecavir, in appropriate clinical situations, for treatment of hepatitis B [e.g. prior intolerance to Tenofovir (TDF), viral resistance to lamivudine (3TC) / Emtricitabine (FTC)] after discussion and agreement between the investigator and the medical monitor.
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of IP.
* Any evidence of primary viral resistance to PIs or INIs based on the presence of any major resistance-associated mutation.
* The subject's virus does not yield results using genotype at Screening (assay data is essential for eligibility determination).
* Any verified Grade 4 laboratory abnormality, with the exception of Grade 4 triglycerides. A single repeat test is allowed during the Screening period to verify a result.
* Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound.
* Alanine aminotransferase (ALT) >=5 times the upper limit of normal (ULN) or ALT >=3xULN and bilirubin >=1.5xULN (with >35% direct bilirubin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (50):
- Argentina (5):
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
- Brazil (4):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, São Paulo, São Paulo
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Chile (3):
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- China (3):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
- GSK Investigational Site, Bogotá, Colombia
- GSK Investigational Site, Nairobi, Kenya
- Mexico (4):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Distrito Federal
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- Peru (2):
  - GSK Investigational Site, Callao
  - GSK Investigational Site, Lima
- Romania (4):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Târgu Mureş
- Russia (9):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Toliyatti
  - GSK Investigational Site, Yekaterinburg
- South Africa (5):
  - GSK Investigational Site, Soweto, Gauteng
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Observatory, Cape Town
  - GSK Investigational Site, Westdene
- Thailand (5):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Nonthaburi
  - GSK Investigational Site, Ratchatewi
- Ukraine (4):
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on ViiV's data sharing criteria can be found at: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/

REFERENCES:
- [Background] Aboud M, Kaplan R, Lombaard J, Zhang F, Hidalgo JA, Mamedova E, Losso MH, Chetchotisakd P, Brites C, Sievers J, Brown D, Hopking J, Underwood M, Nascimento MC, Punekar Y, Gartland M, Smith K. Dolutegravir versus ritonavir-boosted lopinavir both with dual nucleoside reverse transcriptase inhibitor therapy in adults with HIV-1 infection in whom first-line therapy has failed (DAWNING): an open-label, non-inferiority, phase 3b trial. Lancet Infect Dis. 2019 Mar;19(3):253-264. doi: 10.1016/S1473-3099(19)30036-2. Epub 2019 Feb 4. PMID 30732940
- [Background] Underwood M, Horton J, Nangle K, Hopking J, Smith K, Aboud M, Wynne B, Sievers J, Stewart EL, Wang R. Integrase Inhibitor Resistance Mechanisms and Structural Characteristics in Antiretroviral Therapy-Experienced, Integrase Inhibitor-Naive Adults with HIV-1 Infection Treated with Dolutegravir plus Two Nucleoside Reverse Transcriptase Inhibitors in the DAWNING Study. Antimicrob Agents Chemother. 2022 Jan 18;66(1):e0164321. doi: 10.1128/AAC.01643-21. Epub 2021 Oct 25. PMID 34694877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study assessed antiviral activity and safety of dolutegravir (DTG) in human immunodeficiency virus-1 (HIV-1) infected participants with treatment failure on first line therapy. The study consisted of Randomized Phase followed by Continuation Phase.
Pre-assignment Details: A total of 627 participants were randomized in 1:1 to receive DTG or lopinavir/ritonavir (LPV/RTV). Three participants in the LPV/RTV group were randomized but not treated. A total of 624 participants received at least one dose of study medication creating the intent to treat-exposed (ITT-E) Population.
Groups:
- Participants Receiving DTG-Randomized Phase: Participants received 1 tablet of 50 milligrams (mg) of DTG once daily along with 2 Nucleoside reverse transcriptase inhibitors (NRTIs) via oral route for 52 weeks during Randomized Phase.
- Participants Receiving LPV/RTV-Randomized Phase: Participants received 4 tablets containing 200/50 mg of LPV/RTV once daily or 2 tablets containing 200/50 mg of LPV/RTV twice daily along with 2 NRTIs via oral route for 52 weeks during Randomized Phase.
- Participants Receiving DTG-Continuation Phase: Participants received DTG in the Continuation Phase until it was either locally approved or commercial supplies were available.
Period: Randomized Phase (Up to Week 52)
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase | Participants Receiving DTG-Continuation Phase
Started (Randomized) | 312 | 315 | 0
ITT-E Population | 312 | 312 | 0
Completed | 275 | 245 | 0
Not Completed | 37 | 70 | 0
Not completed — Reached stopping criteria | 0 | 1 | 0
Not completed — Adverse Event | 8 | 18 | 0
Not completed — Lack of Efficacy | 10 | 22 | 0
Not completed — Protocol Violation | 7 | 8 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 0
Not completed — Physician Decision | 0 | 9 | 0
Not completed — Lost to Follow-up | 7 | 5 | 0
Not completed — Randomized, but did not receive treatment | 0 | 3 | 0
Period: Continuation Phase(From Weeks 52 to 295)
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase | Participants Receiving DTG-Continuation Phase
Started | 0 | 0 | 274 (274 participants from the Randomized entered in the Continuation Phase.)
Completed | 0 | 0 | 225
Not Completed | 0 | 0 | 49
Not completed — Adverse Event | 0 | 0 | 8
Not completed — Lack of Efficacy | 0 | 0 | 16
Not completed — Protocol Violation | 0 | 0 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 6
Not completed — Physician Decision | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: Baseline Characteristic data are reported for members of the ITT-E Population which comprised of all participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase | Total
Number analyzed (Participants) | 312 | 312 | 624
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.5 (9.13) | 38.7 (9.35) | 38.1 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 103 | 219
  Male | 196 | 209 | 405
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, customized: American Indian or Alaska native | 42 | 53 | 95
  Race, customized: Asian- Central/South Asian Heritage | 1 | 0 | 1
  Race, customized: Asian - East Asian Heritage | 21 | 31 | 52
  Race, customized: Asian - South East Asian Heritage | 28 | 25 | 53
  Race, customized: White - Arabic/North African Heritage | 2 | 0 | 2
  Race, customized: White - White/Caucasian/European Heritage | 88 | 90 | 178
  Race, customized: Mixed White Race | 0 | 1 | 1
  Race, customized: Black or African American Heritage | 130 | 112 | 242

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) <50 Copies Per Milliliter (c/mL) at Week 48
Description: Percentage of participants with plasma HIV 1 RNA <50 c/mL at Week 48 using the Food and Drug Administration (FDA) snapshot algorithm was assessed to demonstrate the non-inferior activity of DTG plus 2 NRTI's compared to LPV/RTV plus 2 NRTI's. Analysis was performed on Intent-to-treat exposed (ITT-E) Population, which comprised of all randomized participants who received at least one dose of study medication. Percentage values are rounded off.
Time Frame: Week 48
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 312 | 312
Percentage of participants | 84 | 70
Statistical Analysis 1: Comparison: Participants Receiving DTG-Randomized Phase vs Participants Receiving LPV/RTV-Randomized Phase; Test type: Superiority — Non-inferiority of DTG plus 2 NRTI's was to be declared if the lower bound of 95% confidence interval (CI) for the difference in snapshot response rates (DTG - LPV/RTV) is greater than - 12%. This was also performed using the Per-Protocol (PP) Population. If both analyses show non-inferiority, the hypothesis of antiviral effect of DTG + 2 NRTI's was superior to LPV/RTV + 2 NRTIs was to be tested; p < .001, Cochran-Mantel-Haenszel; Proportion difference = 13.8, 95% CI 2-sided [7.3 to 20.3] — Adjusted proportion difference, calculated as proportion on DTG minus that on LPV/RTV and based on Cochran-Mantel Haenszel stratified analysis adjusting for Baseline plasma HIV-1 RNA and number of fully active background NRTIs, has been presented; Superiority would be declared if the lower end of the confidence interval was above 0%

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 24
Description: Percentage of participants with plasma HIV 1 RNA <50 c/mL at Week 24 using the FDA snapshot algorithm was assessed to demonstrate the non-inferior activity of DTG plus 2 NRTI's compared to LPV/RTV plus 2 NRTI's. Percentage values are rounded off.
Time Frame: Week 24
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 312 | 312
Percentage of participants | 82 | 69

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <400 c/mL at Weeks 24 and 48
Description: Percentage of participants with plasma HIV 1 RNA <400 c/mL at Week 24 and 48 using the FDA snapshot algorithm were evaluated. Percentage values are rounded off.
Time Frame: Week 24 and Week 48
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 312 | 312
Percentage of participants
  Week 24 | 90 | 84
  Week 48 | 88 | 77

4. Secondary Outcome: Percentage of Participants Without Virologic or Tolerability Failure at Week 24 and Week 48
Description: Virologic or tolerability failure was defined as treatment-related discontinuation (meeting confirmed virologic withdrawal criteria, treatment-related adverse event, safety stopping criteria, and lack of efficacy). Percentage of participants without virologic failure by Week 24 and Week 48 have been presented. Participants who did not met the protocol defined confirmed virologic withdrawal criteria and are ongoing in the study, or who had discontinued for non-treatment related reasons were censored.
Time Frame: Week 24 and Week 48
Population: ITT-E Population
Measure: Number; unit: Percentage of participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 312 | 312
Percentage of participants
  Week 24 | 97.6 | 91.9
  Week 48 | 96.0 | 86.1
Statistical Analysis 1: Comparison: Participants Receiving DTG-Randomized Phase vs Participants Receiving LPV/RTV-Randomized Phase; Test type: Other; Proportion difference = 5.7, 95% CI 2-sided [2.2 to 9.3] — Proportion difference, calculated as proportion on DTG minus proportion on LPV/RTV, at Week 24 has been presented
Statistical Analysis 2: Comparison: Participants Receiving DTG-Randomized Phase vs Participants Receiving LPV/RTV-Randomized Phase; Test type: Other; Proportion difference = 9.8, 95% CI 2-sided [5.3 to 14.4] — Proportion difference, calculated as proportion on DTG minus proportion on LPV/RTV, at Week 48 has been presented

5. Secondary Outcome: Time to Viral Suppression at Week 48
Description: Viral suppression was defined as HIV-1 RNA <50 c/mL. Time to viral suppression was analyzed and median and interquartile range has been presented.
Time Frame: Week 48
Population: ITT-E Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 312 | 312
Days | 29.0 [29.0 to 57.0] | 111.0 [35.0 to 167.0]

6. Secondary Outcome: Change From Baseline in Helper-inducer T-lymphocyte Having Surface Antigen Cluster of Differentiation (CD4+) Cell Count at Weeks 24 and 48
Description: Blood was collected and CD4+ cell count assessment was carried out at indicated time points to evaluate the immunological activity of DTG compared to LPV/RTV. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Week 24 and Week 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Median (Inter-Quartile Range); unit: Cells per cubic millimeter (Cells/mm^3)
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 312 | 312
Cells per cubic millimeter (Cells/mm^3)
  Week 24; n= 291, 285: number analyzed (Participants) | 291 | 285
  Week 24; n= 291, 285 | 84.0 [31.0 to 146.0] | 82.0 [31.0 to 146.0]
  Week 48; n= 275, 251: number analyzed (Participants) | 275 | 251
  Week 48; n= 275, 251 | 120.0 [63.0 to 204.0] | 118.0 [66.0 to 191.0]

7. Secondary Outcome: Number of Participants With Disease Progression-Randomized + Continuation Phase
Description: Disease progression included HIV-associated conditions, acquired immune deficiency syndrome (AIDS) and death. Number of participants with disease progression to Centers for Disease Control and Prevention (CDC) class C or death have been presented.
Time Frame: Up to Week 348
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Groups:
- DTG in Randomized Phase Followed by Continuation Phase: Participants received 1 tablet of 50 mg of DTG once daily along with 2 NRTIs via oral route for 52 weeks during Randomized Phase. Participants who completed 52 weeks of treatment, continued to receive DTG in the Continuation Phase until it was either locally approved or commercial supplies were available.
- LPV/RTV-Randomized Phase Followed by DTG in Continuation Phase: Participants received 4 tablets containing 200/50 mg of LPV/RTV once daily or 2 tablets containing 200/50 mg of LPV/RTV twice daily along with 2 NRTIs via oral route for 52 weeks during Randomized Phase. Participants switched to DTG by Week 52 continued to receive DTG in Continuation Phase until it was either locally approved and commercial supplies were available.
Arm/Group | DTG in Randomized Phase Followed by Continuation Phase | LPV/RTV-Randomized Phase Followed by DTG in Continuation Phase
Number analyzed (Participants) | 312 | 312
Participants | 10 | 7

8. Secondary Outcome: Number of Participants With Treatment-emergent Genotypic Resistance-Randomized Phase
Description: Number of participants, who met confirmed virologic withdrawal (CVW) criteria with paired Baseline and time of CVW resistance data with treatment emergent genotypic resistance to Integrase strand transfer inhibitor (INSTI), NRTI, Protease inhibitor (PI) were summarized. Viral Genotypic Population comprised of all participants in the ITT-E population with available On-treatment genotypic resistance data at the time confirmed virologic withdrawal criterion was met during Randomized Phase.
Time Frame: Up to Week 52
Population: Viral genotypic Population. Only those participants with data available at specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 11 | 30
Participants
  INSTI | 3 | 0
  NRTI | 1 | 3
  PI | 0 | 0

9. Secondary Outcome: Number of Participants With Treatment-emergent Genotypic Resistance-Continuation Phase
Description: Number of participants, who met confirmed virologic withdrawal criteria with paired Baseline and time of CVW resistance data, with treatment emergent genotypic resistance to Integrase strand transfer inhibitor (INSTI), NRTI, Protease inhibitor (PI) were summarized. Analysis was performed on Viral Genotypic Continuation Population which comprised all participants in the ITT-E- Continuation Population with available on-treatment genotypic resistance data in the Continuation Phase.
Time Frame: Up to Week 295
Population: Viral genotypic continuation Population. Only those participants with data available at specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG-Continuation Phase
Number analyzed (Participants) | 16
Participants
  INSTI | 5
  NRTI | 2
  PI | 0

10. Secondary Outcome: Number of Participants With Fold Change in Treatment-emergent Phenotypic Resistance From Baseline-Randomized Phase
Description: Number of participants with fold change in treatment-emergent phenotypic resistance from Baseline to DTG, LPV/RTV was counted to assess the development of viral resistance. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-dose visit value minus Baseline value. Change in grade 0 to >2 from Baseline is presented. Analysis was performed on viral phenotypic Population, which comprised of all participants in the ITT-E Population with available On-treatment phenotypic resistance data at the time confirmed virologic withdrawal criterion is met during Randomized Phase.
Time Frame: Baseline (Day 1, Pre-dose) and up to Week 52
Population: Viral Phenotypic Population. Only those participants with data available at specified time point were analyzed (represented by n=X) in category titles.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 11 | 29
Participants
  DTG; <1; n=11, 23: number analyzed (Participants) | 11 | 23
  DTG; <1; n=11, 23 | 5 | 18
  DTG; 1-<2; n=11, 23: number analyzed (Participants) | 11 | 23
  DTG; 1-<2; n=11, 23 | 2 | 5
  DTG; 2-<4; n=11, 23: number analyzed (Participants) | 11 | 23
  DTG; 2-<4; n=11, 23 | 1 | 0
  DTG; 4-<8; n=11, 23: number analyzed (Participants) | 11 | 23
  DTG; 4-<8; n=11, 23 | 0 | 0
  DTG; >=8; n=11, 23: number analyzed (Participants) | 11 | 23
  DTG; >=8; n=11, 23 | 3 | 0
  LPV/RTV; <1; n=11, 29 | 7 | 21
  LPV/RTV; 1-<2; n=11, 29 | 4 | 8
  LPV/RTV; 2-<4; n=11, 29 | 0 | 0
  LPV/RTV; 4-<8; n=11, 29 | 0 | 0
  LPV/RTV; >=8; n=11, 29 | 0 | 0

11. Secondary Outcome: Number of Participants With Fold Change in Treatment-emergent Phenotypic Resistance From Baseline-Continuation Phase
Description: Number of participants with fold change in treatment-emergent phenotypic resistance from Baseline to DTG was counted to assess the development of viral resistance. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-dose visit value minus Baseline value. Change in grade 0 to >2 from Baseline is presented. Analysis was performed on Viral Phenotypic Continuation Population which comprises all participants in the ITT-E- Continuation Population with available on-treatment phenotypic resistance data in the Continuation Phase.
Time Frame: Baseline (Day 1, Pre-dose) and up to Week 295
Population: Viral Phenotypic continuation Population. Only those participants with data available at specified time point were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Receiving DTG in Continuation Phase: Participants received DTG in the Continuation Phase until it was either locally approved or commercial supplies were available.
Arm/Group | Participants Receiving DTG in Continuation Phase
Number analyzed (Participants) | 15
Participants
  DTG; <1 | 8
  DTG; 1-<2 | 3
  DTG; 2-<4 | 0
  DTG; 4-<8 | 0
  DTG; >=8 | 4

12. Secondary Outcome: Number of Participants With Non-serious Adverse Events (AEs) With >=2% Frequency Threshold and Serious Adverse Events (SAEs)-Randomized Phase
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, other situations as per medical or scientific judgment and is associated with liver injury or impaired liver function. Safety Population was used which comprised of all participants who received at least one dose of study treatment. Adverse events which were not Serious were considered as Non-Serious adverse events.
Time Frame: Up to Week 52
Population: Safety Population. Two participants who were randomized to receive LPV/RTV, received DTG and were included in DTG group for Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Participants
  Any non-serious AEs | 155 | 202
  Any SAEs | 20 | 20

13. Secondary Outcome: Number of Participants With Non-serious AEs With >=2% Frequency Threshold and SAEs-Continuation Phase
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, other situations as per medical or scientific judgment and is associated with liver injury or impaired liver function. Adverse events which were not Serious were considered as non-serious AEs.
Time Frame: Up to Week 295
Population: Safety-Continuation Population comprised all participants in the Safety Population who received at least one dose of Investigational Product after entering the Continuation Phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG-Continuation Phase
Number analyzed (Participants) | 274
Participants
  Any non-serious AEs | 150
  Any SAEs | 29

14. Secondary Outcome: Number of Participants With Non-serious AEs With >=2% Frequency Threshold and SAEs-Randomized + Continuation Phase
Description: as for outcome 13
Time Frame: Up to Week 348
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Groups:
- DTG- Randomized Phase Followed by Continuation Phase: Participants received 1 tablet of 50 mg of DTG once daily along with 2 NRTIs via oral route for 52 weeks during Randomized Phase. Participants who completed 52 weeks of treatment, continued to receive DTG in the Continuation Phase until it was either locally approved or commercial supplies were available.
- LPV/RTV- Randomized Phase Followed by DTG-Continuation Phase: Participants received 4 tablets containing 200/50 mg of LPV/RTV once daily or 2 tablets containing 200/50 mg of LPV/RTV twice daily along with 2 NRTIs via oral route for 52 weeks during Randomized Phase. Participants switched to DTG by Week 52 continued to receive DTG in Continuation Phase until it was either locally approved and commercial supplies were available.
Arm/Group | DTG- Randomized Phase Followed by Continuation Phase | LPV/RTV- Randomized Phase Followed by DTG-Continuation Phase
Number analyzed (Participants) | 314 | 310
Participants
  Any non-serious AEs | 218 | 213
  Any SAEs | 47 | 20

15. Secondary Outcome: Change From Baseline in Glucose, Chloride, Carbon-di-oxide (CO2), Potassium, Phosphate, Sodium, Urea, Cholesterol, High Density Lipoprotein (HDL) Cholesterol, Low Density Lipoprotein (LDL) Cholesterol and Triglycerides
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including glucose, chloride, carbon-di-oxide (CO2), potassium, phosphate, sodium, urea, cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol and triglycerides. Lipid parameters were evaluated in fasting condition. Change from Baseline in clinical chemistry parameters at Weeks 4, 8, 16, 24, 36, 48, 52 are presented. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 8, Week 16, Week 24, Week 36, Week 48 and Week 52
Population: Safety Population. Two participants who were randomized to receive LPV/RTV, received DTG and were included in DTG group for Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Millimoles per liter
  Glucose; Week 4; n= 279, 277: number analyzed (Participants) | 279 | 277
  Glucose; Week 4; n= 279, 277 | 0.07 (0.789) | 0.01 (0.661)
  Glucose; Week 8; n= 273, 271: number analyzed (Participants) | 273 | 271
  Glucose; Week 8; n= 273, 271 | 0.08 (1.086) | -0.00 (0.914)
  Glucose; Week 16; n= 280, 275: number analyzed (Participants) | 280 | 275
  Glucose; Week 16; n= 280, 275 | 0.07 (0.740) | -0.06 (1.060)
  Glucose; Week 24; n= 288, 276: number analyzed (Participants) | 288 | 276
  Glucose; Week 24; n= 288, 276 | 0.22 (2.286) | -0.04 (1.037)
  Glucose; Week 36; n= 270, 257: number analyzed (Participants) | 270 | 257
  Glucose; Week 36; n= 270, 257 | 0.18 (1.056) | -0.01 (1.176)
  Glucose; Week 48; n= 269, 237: number analyzed (Participants) | 269 | 237
  Glucose; Week 48; n= 269, 237 | 0.12 (1.099) | -0.01 (1.028)
  Glucose; Week 52; n= 258, 221: number analyzed (Participants) | 258 | 221
  Glucose; Week 52; n= 258, 221 | 0.16 (1.142) | -0.01 (1.443)
  Chloride; Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  Chloride; Week 4; n= 306, 302 | -0.20 (2.692) | -0.96 (2.751)
  Chloride; Week 8; n= 301, 298: number analyzed (Participants) | 301 | 298
  Chloride; Week 8; n= 301, 298 | -0.15 (2.752) | -1.00 (2.833)
  Chloride; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  Chloride; Week 16; n= 294, 292 | 0.04 (2.709) | -0.78 (2.773)
  Chloride; Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  Chloride; Week 24; n= 295, 286 | -0.17 (2.887) | -0.67 (2.818)
  Chloride; Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  Chloride; Week 36; n= 289, 276 | -0.18 (2.569) | -0.51 (2.880)
  Chloride; Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  Chloride; Week 48; n= 278, 247 | -0.03 (2.663) | -0.81 (2.441)
  Chloride; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  Chloride; Week 52; n= 276, 238 | 0.06 (3.111) | -0.38 (2.739)
  CO2; Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  CO2; Week 4; n= 306, 302 | 0.12 (2.754) | -0.22 (2.650)
  CO2; Week 8; n= 301, 297: number analyzed (Participants) | 301 | 297
  CO2; Week 8; n= 301, 297 | -0.01 (2.695) | -0.09 (2.564)
  CO2; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  CO2; Week 16; n= 294, 292 | 0.21 (2.978) | 0.04 (2.638)
  CO2; Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  CO2; Week 24; n= 295, 286 | 0.13 (2.818) | -0.08 (2.777)
  CO2; Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  CO2; Week 36; n= 289, 276 | 0.16 (2.620) | -0.12 (2.861)
  CO2; Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  CO2; Week 48; n= 278, 247 | 0.06 (2.672) | 0.28 (2.867)
  CO2; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  CO2; Week 52; n= 276, 238 | 0.04 (2.736) | 0.12 (2.555)
  Potassium; Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  Potassium; Week 4; n= 306, 302 | 0.07 (0.373) | -0.02 (0.432)
  Potassium; Week 8; n= 301, 297: number analyzed (Participants) | 301 | 297
  Potassium; Week 8; n= 301, 297 | 0.09 (0.350) | 0.00 (0.428)
  Potassium; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  Potassium; Week 16; n= 294, 292 | 0.10 (0.375) | 0.03 (0.443)
  Potassium; Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  Potassium; Week 24; n= 295, 286 | 0.11 (0.401) | 0.03 (0.433)
  Potassium; Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  Potassium; Week 36; n= 289, 276 | 0.08 (0.363) | -0.03 (0.417)
  Potassium; Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  Potassium; Week 48; n= 278, 247 | 0.07 (0.369) | 0.05 (0.423)
  Potassium; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  Potassium; Week 52; n= 276, 238 | 0.11 (0.412) | 0.04 (0.416)
  Phosphate; Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  Phosphate; Week 4; n= 306, 302 | 0.11 (0.188) | 0.01 (0.206)
  Phosphate; Week 8; n= 301, 298: number analyzed (Participants) | 301 | 298
  Phosphate; Week 8; n= 301, 298 | 0.11 (0.182) | 0.03 (0.187)
  Phosphate; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  Phosphate; Week 16; n= 294, 292 | 0.10 (0.180) | 0.03 (0.193)
  Phosphate; Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  Phosphate; Week 24; n= 295, 286 | 0.11 (0.174) | 0.03 (0.200)
  Phosphate; Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  Phosphate; Week 36; n= 289, 276 | 0.08 (0.196) | 0.01 (0.217)
  Phosphate; Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  Phosphate; Week 48; n= 278, 247 | 0.06 (0.193) | 0.03 (0.209)
  Phosphate; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  Phosphate; Week 52; n= 276, 238 | 0.06 (0.203) | 0.01 (0.197)
  Sodium; Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  Sodium; Week 4; n= 306, 302 | -0.20 (2.393) | -0.80 (2.284)
  Sodium; Week 8; n= 301, 298: number analyzed (Participants) | 301 | 298
  Sodium; Week 8; n= 301, 298 | -0.12 (2.420) | -0.87 (2.569)
  Sodium; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  Sodium; Week 16; n= 294, 292 | 0.29 (2.364) | -0.58 (2.449)
  Sodium; Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  Sodium; Week 24; n= 295, 286 | -0.07 (2.472) | -0.53 (2.446)
  Sodium; Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  Sodium; Week 36; n= 289, 276 | 0.08 (2.375) | -0.51 (2.410)
  Sodium; Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  Sodium; Week 48; n= 278, 247 | 0.22 (2.277) | -0.62 (2.505)
  Sodium; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  Sodium; Week 52; n= 276, 238 | 0.09 (2.886) | -0.37 (2.402)
  Urea; Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  Urea; Week 4; n= 306, 302 | 0.21 (1.658) | 0.18 (1.253)
  Urea; Week 8; n= 301, 298: number analyzed (Participants) | 301 | 298
  Urea; Week 8; n= 301, 298 | 0.21 (1.214) | 0.23 (1.205)
  Urea; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  Urea; Week 16; n= 294, 292 | 0.25 (1.269) | 0.29 (1.344)
  Urea; Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  Urea; Week 24; n= 295, 286 | 0.35 (1.236) | 0.17 (1.308)
  Urea; Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  Urea; Week 36; n= 289, 276 | 0.11 (1.165) | 0.20 (1.284)
  Urea; Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  Urea; Week 48; n= 278, 247 | 0.19 (1.260) | 0.18 (1.241)
  Urea; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  Urea; Week 52; n= 276, 238 | 0.30 (1.482) | 0.32 (1.311)
  Cholesterol; Week 4; n= 4, 6: number analyzed (Participants) | 4 | 6
  Cholesterol; Week 4; n= 4, 6 | -0.88 (1.081) | 1.22 (1.963)
  Cholesterol; Week 8; n= 7, 10: number analyzed (Participants) | 7 | 10
  Cholesterol; Week 8; n= 7, 10 | -0.37 (1.158) | 1.04 (1.577)
  Cholesterol; Week 16; n= 270, 261: number analyzed (Participants) | 270 | 261
  Cholesterol; Week 16; n= 270, 261 | -0.22 (0.878) | 0.31 (0.872)
  Cholesterol; Week 24; n= 280, 271: number analyzed (Participants) | 280 | 271
  Cholesterol; Week 24; n= 280, 271 | -0.23 (0.760) | 0.29 (0.934)
  Cholesterol; Week 36; n= 283, 272: number analyzed (Participants) | 283 | 272
  Cholesterol; Week 36; n= 283, 272 | -0.24 (0.789) | 0.28 (0.901)
  Cholesterol; Week 48; n= 276, 272: number analyzed (Participants) | 276 | 272
  Cholesterol; Week 48; n= 276, 272 | -0.10 (0.808) | 0.38 (0.946)
  Cholesterol; Week 52; n= 7, 6: number analyzed (Participants) | 7 | 6
  Cholesterol; Week 52; n= 7, 6 | 0.35 (0.593) | -0.18 (0.850)
  HDL cholesterol; Week 4; n= 4, 6: number analyzed (Participants) | 4 | 6
  HDL cholesterol; Week 4; n= 4, 6 | -0.18 (0.197) | 0.10 (0.191)
  HDL cholesterol; Week 8; n= 7,10: number analyzed (Participants) | 7 | 10
  HDL cholesterol; Week 8; n= 7,10 | -0.01 (0.262) | 0.08 (0.363)
  HDL cholesterol; Week 16; n= 270, 261: number analyzed (Participants) | 270 | 261
  HDL cholesterol; Week 16; n= 270, 261 | -0.02 (0.300) | -0.00 (0.341)
  HDL cholesterol; Week 24; n= 280, 271: number analyzed (Participants) | 280 | 271
  HDL cholesterol; Week 24; n= 280, 271 | -0.02 (0.319) | 0.00 (0.339)
  HDL cholesterol; Week 36; n= 283, 272: number analyzed (Participants) | 283 | 272
  HDL cholesterol; Week 36; n= 283, 272 | -0.02 (0.319) | 0.00 (0.340)
  HDL cholesterol; Week 48; n= 276, 272: number analyzed (Participants) | 276 | 272
  HDL cholesterol; Week 48; n= 276, 272 | -0.02 (0.298) | 0.03 (0.353)
  HDL cholesterol; Week 52; n= 7,6: number analyzed (Participants) | 7 | 6
  HDL cholesterol; Week 52; n= 7,6 | 0.18 (0.327) | 0.13 (0.327)
  LDL cholesterol; Week 4; n= 4, 3: number analyzed (Participants) | 4 | 3
  LDL cholesterol; Week 4; n= 4, 3 | -0.29 (1.157) | -0.17 (0.398)
  LDL cholesterol; Week 8; n= 7, 8: number analyzed (Participants) | 7 | 8
  LDL cholesterol; Week 8; n= 7, 8 | -0.09 (0.911) | 0.50 (0.720)
  LDL cholesterol; Week 16; n= 259, 246: number analyzed (Participants) | 259 | 246
  LDL cholesterol; Week 16; n= 259, 246 | -0.10 (0.674) | 0.06 (0.644)
  LDL cholesterol; Week 24; n= 272, 261: number analyzed (Participants) | 272 | 261
  LDL cholesterol; Week 24; n= 272, 261 | -0.10 (0.601) | 0.05 (0.652)
  LDL cholesterol; Week 36; n= 274, 261: number analyzed (Participants) | 274 | 261
  LDL cholesterol; Week 36; n= 274, 261 | -0.11 (0.606) | 0.05 (0.659)
  LDL cholesterol; Week 48; n= 269, 264: number analyzed (Participants) | 269 | 264
  LDL cholesterol; Week 48; n= 269, 264 | -0.01 (0.633) | 0.11 (0.682)
  LDL cholesterol; Week 52; n= 7, 6: number analyzed (Participants) | 7 | 6
  LDL cholesterol; Week 52; n= 7, 6 | 0.06 (0.511) | -0.25 (0.857)
  Triglycerides; Week 4; n= 4, 6: number analyzed (Participants) | 4 | 6
  Triglycerides; Week 4; n= 4, 6 | -0.89 (0.852) | 4.23 (5.773)
  Triglycerides; Week 8; n= 7, 10: number analyzed (Participants) | 7 | 10
  Triglycerides; Week 8; n= 7, 10 | -0.57 (1.153) | 1.95 (5.131)
  Triglycerides; Week 16; n= 270, 261: number analyzed (Participants) | 270 | 261
  Triglycerides; Week 16; n= 270, 261 | -0.32 (1.131) | 0.63 (1.289)
  Triglycerides; Week 24; n= 280, 271: number analyzed (Participants) | 280 | 271
  Triglycerides; Week 24; n= 280, 271 | -0.32 (0.997) | 0.67 (1.826)
  Triglycerides; Week 36; n= 283, 272: number analyzed (Participants) | 283 | 272
  Triglycerides; Week 36; n= 283, 272 | -0.31 (1.289) | 0.61 (1.497)
  Triglycerides; Week 48; n= 276, 272: number analyzed (Participants) | 276 | 272
  Triglycerides; Week 48; n= 276, 272 | -0.24 (1.120) | 0.57 (1.488)
  Triglycerides; Week 52; n= 7, 6: number analyzed (Participants) | 7 | 6
  Triglycerides; Week 52; n= 7, 6 | 0.22 (0.769) | -0.15 (0.259)

16. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatine Kinase Values
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including ALP, ALT, AST and creatine kinase. Change from Baseline in clinical chemistry parameters at Weeks 4, 8, 16, 24, 36, 48, 52 are presented. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 8, Week 16, Week 24, Week 36, Week 48 and Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: International unit per liter
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
International unit per liter
  ALP; Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  ALP; Week 4; n= 306, 302 | -12.24 (21.900) | -14.94 (22.979)
  ALP; Week 8; n= 301, 298: number analyzed (Participants) | 301 | 298
  ALP; Week 8; n= 301, 298 | -13.73 (26.135) | -13.46 (29.998)
  ALP; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  ALP; Week 16; n= 294, 292 | -13.87 (31.452) | -11.38 (26.190)
  ALP; Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  ALP; Week 24; n= 295, 286 | -14.19 (27.800) | -6.06 (50.943)
  ALP; Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  ALP; Week 36; n= 289, 276 | -13.53 (28.875) | -7.85 (30.394)
  ALP; Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  ALP; Week 48; n= 278, 247 | -14.10 (28.935) | -6.87 (32.071)
  ALP; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  ALP; Week 52; n= 276, 238 | -13.81 (29.317) | -7.23 (31.046)
  ALT; Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  ALT; Week 4; n= 306, 302 | -2.50 (17.285) | -10.25 (17.639)
  ALT; Week 8; n= 301, 298: number analyzed (Participants) | 301 | 298
  ALT; Week 8; n= 301, 298 | -2.49 (19.222) | -9.04 (25.556)
  ALT; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  ALT; Week 16; n= 294, 292 | -4.32 (18.502) | -8.59 (24.507)
  ALT; Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  ALT; Week 24; n= 295, 286 | -3.87 (20.108) | -9.20 (33.054)
  ALT; Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  ALT; Week 36; n= 289, 276 | -1.31 (25.356) | -11.16 (22.196)
  ALT; Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  ALT; Week 48; n= 278, 247 | 0.19 (39.985) | -6.47 (51.492)
  ALT; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  ALT; Week 52; n= 276, 238 | -1.04 (23.232) | -10.63 (25.508)
  AST; Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  AST; Week 4; n= 306, 302 | -3.56 (17.463) | -7.68 (13.654)
  AST; Week 8; n= 301, 297: number analyzed (Participants) | 301 | 297
  AST; Week 8; n= 301, 297 | -2.89 (17.934) | -6.64 (21.295)
  AST; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  AST; Week 16; n= 294, 292 | -4.70 (17.445) | -6.49 (18.143)
  AST; Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  AST; Week 24; n= 295, 286 | -3.83 (17.713) | -6.45 (28.933)
  AST; Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  AST; Week 36; n= 289, 276 | -1.76 (22.437) | -8.36 (21.550)
  AST; Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  AST; Week 48; n= 278, 247 | -2.03 (28.194) | -6.43 (27.155)
  AST; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  AST; Week 52; n= 276, 238 | -1.51 (22.645) | -7.55 (28.125)
  Creatine kinase; Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  Creatine kinase; Week 4; n= 306, 302 | -2.85 (215.820) | -15.59 (106.738)
  Creatine kinase; Week 8; n= 301, 298: number analyzed (Participants) | 301 | 298
  Creatine kinase; Week 8; n= 301, 298 | 18.61 (312.940) | -10.42 (128.109)
  Creatine kinase; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  Creatine kinase; Week 16; n= 294, 292 | 11.75 (180.905) | 11.62 (203.660)
  Creatine kinase; Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  Creatine kinase; Week 24; n= 295, 286 | 34.71 (312.173) | -0.28 (186.927)
  Creatine kinase; Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  Creatine kinase; Week 36; n= 289, 276 | 72.34 (892.830) | -5.08 (135.191)
  Creatine kinase; Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  Creatine kinase; Week 48; n= 278, 247 | 45.50 (451.135) | 16.52 (295.891)
  Creatine kinase; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  Creatine kinase; Week 52; n= 276, 238 | 39.24 (228.026) | 54.97 (628.621)

17. Secondary Outcome: Change From Baseline in Albumin Values
Description: Blood samples were collected from participants to evaluate clinical chemistry parameter including albumin. Change from Baseline in clinical chemistry parameters at Weeks 4, 8, 16, 24, 36, 48, 52 are presented. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 8, Week 16, Week 24, Week 36, Week 48 and Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Gram per liter
  Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  Week 4; n= 306, 302 | -0.39 (2.554) | -0.51 (2.670)
  Week 8; n= 301, 298: number analyzed (Participants) | 301 | 298
  Week 8; n= 301, 298 | 0.09 (2.792) | -0.67 (2.828)
  Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  Week 16; n= 294, 292 | 0.50 (3.148) | -0.28 (3.062)
  Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  Week 24; n= 295, 286 | 0.63 (3.326) | -0.06 (3.207)
  Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  Week 36; n= 289, 276 | 0.76 (3.479) | -0.11 (3.091)
  Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  Week 48; n= 278, 247 | 0.71 (3.250) | 0.11 (2.912)
  Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  Week 52; n= 276, 238 | 0.83 (3.605) | -0.15 (3.142)

18. Secondary Outcome: Change From Baseline in Creatinine and Bilirubin Values
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including creatinine and bilirubin. Change from Baseline in clinical chemistry parameters at Weeks 4, 8, 16, 24, 36, 48, 52 are presented. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 8, Week 16, Week 24, Week 36, Week 48 and Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Micromoles per liter
  Creatinine; Week 4; n= 306, 302: number analyzed (Participants) | 306 | 302
  Creatinine; Week 4; n= 306, 302 | 9.68 (9.308) | 4.69 (8.575)
  Creatinine; Week 8; n= 301, 298: number analyzed (Participants) | 301 | 298
  Creatinine; Week 8; n= 301, 298 | 10.81 (8.414) | 5.57 (9.214)
  Creatinine; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  Creatinine; Week 16; n= 294, 292 | 12.46 (9.065) | 5.19 (9.648)
  Creatinine; Week 24; n= 295, 286: number analyzed (Participants) | 295 | 286
  Creatinine; Week 24; n= 295, 286 | 12.96 (10.248) | 5.75 (11.606)
  Creatinine; Week 36; n= 289, 276: number analyzed (Participants) | 289 | 276
  Creatinine; Week 36; n= 289, 276 | 12.08 (9.667) | 5.98 (14.737)
  Creatinine; Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  Creatinine; Week 48; n= 278, 247 | 12.92 (9.412) | 6.15 (13.373)
  Creatinine; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  Creatinine; Week 52; n= 276, 238 | 13.22 (10.229) | 6.15 (12.268)
  Bilirubin; Week 4; n= 305, 301: number analyzed (Participants) | 305 | 301
  Bilirubin; Week 4; n= 305, 301 | 1.74 (4.982) | 3.39 (3.997)
  Bilirubin; Week 8; n= 301, 297: number analyzed (Participants) | 301 | 297
  Bilirubin; Week 8; n= 301, 297 | 2.25 (4.344) | 3.76 (5.291)
  Bilirubin; Week 16; n= 294, 292: number analyzed (Participants) | 294 | 292
  Bilirubin; Week 16; n= 294, 292 | 2.79 (4.547) | 3.97 (4.957)
  Bilirubin; Week 24; n= 295, 285: number analyzed (Participants) | 295 | 285
  Bilirubin; Week 24; n= 295, 285 | 3.28 (4.692) | 4.15 (5.422)
  Bilirubin; Week 36; n= 289, 275: number analyzed (Participants) | 289 | 275
  Bilirubin; Week 36; n= 289, 275 | 3.26 (4.925) | 4.43 (5.447)
  Bilirubin; Week 48; n= 278, 246: number analyzed (Participants) | 278 | 246
  Bilirubin; Week 48; n= 278, 246 | 3.19 (4.288) | 4.82 (5.552)
  Bilirubin; Week 52; n= 276, 238: number analyzed (Participants) | 276 | 238
  Bilirubin; Week 52; n= 276, 238 | 3.54 (5.231) | 4.26 (4.644)

19. Secondary Outcome: Change From Baseline in Lipase Values
Description: Blood samples were collected from participants to evaluate clinical chemistry parameter including lipase. Change from Baseline in lipase at Weeks 4, 8, 16, 24, 36, 48, 52 are presented. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 8, Week 16, Week 24, Week 36, Week 48 and Week 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Unit per liter
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Unit per liter
  Week 4; n= 303, 301: number analyzed (Participants) | 303 | 301
  Week 4; n= 303, 301 | 0.17 (11.082) | 1.52 (15.067)
  Week 8; n= 299, 298: number analyzed (Participants) | 299 | 298
  Week 8; n= 299, 298 | 0.79 (13.422) | 0.58 (10.558)
  Week 16; n= 292, 293: number analyzed (Participants) | 292 | 293
  Week 16; n= 292, 293 | 2.01 (17.174) | 0.94 (11.197)
  Week 24; n= 295, 284: number analyzed (Participants) | 295 | 284
  Week 24; n= 295, 284 | 1.19 (15.984) | 1.14 (13.770)
  Week 36; n= 287, 275: number analyzed (Participants) | 287 | 275
  Week 36; n= 287, 275 | 0.49 (15.089) | 0.11 (11.570)
  Week 48; n= 278, 247: number analyzed (Participants) | 278 | 247
  Week 48; n= 278, 247 | 1.13 (14.673) | 1.68 (12.783)
  Week 52; n= 275, 237: number analyzed (Participants) | 275 | 237
  Week 52; n= 275, 237 | 3.18 (22.215) | 1.59 (11.117)

20. Secondary Outcome: Number of Participants With Clinical Chemistry Toxicities -Randomized Phase
Description: Number of participants with clinical chemistry toxicities has been presented. Toxicities were based on the Division of AIDS (DAIDS) grading system. Grade 1=Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Potentially life-threatening. Higher the grade, more severe the symptoms. Lipids and glucose parameters were summarized on fasting data. Data has been reported for clinical chemistry parameters including serum glucose, ALT, Albumin, ALP, AST, Bilirubin, CO2, Creatine kinase, LDL cholesterol calculation, LDL cholesterol direct, Lipase, Phosphate, Potassium, Sodium, Cholesterol, Creatinine and Serum Triglycerides.
Time Frame: Up to Week 52
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Participants
  Serum glucose; Grade 1 | 32 | 27
  Serum glucose; Grade 2 | 10 | 15
  Serum glucose; Grade 3 | 4 | 1
  Serum glucose; Grade 4 | 1 | 0
  ALT; Grade 1 | 27 | 13
  ALT; Grade 2 | 9 | 6
  ALT; Grade 3 | 3 | 2
  ALT; Grade 4 | 1 | 0
  Albumin; Grade 1 | 7 | 3
  Albumin; Grade 2 | 4 | 0
  Albumin; Grade 3 | 0 | 0
  Albumin; Grade 4 | 0 | 0
  ALP; Grade 1 | 9 | 22
  ALP; Grade 2 | 4 | 1
  ALP; Grade 3 | 0 | 1
  ALP; Grade 4 | 0 | 0
  AST; Grade 1 | 29 | 18
  AST; Grade 2 | 10 | 4
  AST; Grade 3 | 2 | 5
  AST; Grade 4 | 1 | 0
  Bilirubin; Grade 1 | 14 | 21
  Bilirubin; Grade 2 | 3 | 11
  Bilirubin; Grade 3 | 2 | 0
  Bilirubin; Grade 4 | 0 | 0
  CO2; Grade 1 | 99 | 105
  CO2; Grade 2 | 24 | 13
  CO2; Grade 3 | 1 | 0
  CO2; Grade 4 | 0 | 0
  Creatine kinase; Grade 1 | 13 | 6
  Creatine kinase; Grade 2 | 2 | 3
  Creatine kinase; Grade 3 | 5 | 3
  Creatine kinase; Grade 4 | 3 | 1
  LDL cholesterol calculation; Grade 1 | 17 | 20
  LDL cholesterol calculation; Grade 2 | 4 | 16
  LDL cholesterol calculation; Grade 3 | 1 | 4
  LDL cholesterol calculation; Grade 4 | 0 | 0
  LDL cholesterol direct; Grade 1 | 3 | 8
  LDL cholesterol direct; Grade 2 | 2 | 4
  LDL cholesterol direct; Grade 3 | 0 | 1
  LDL cholesterol direct; Grade 4 | 0 | 0
  Lipase; Grade 1 | 16 | 12
  Lipase; Grade 2 | 6 | 5
  Lipase; Grade 3 | 1 | 1
  Lipase; Grade 4 | 2 | 0
  Phosphate; Grade 1 | 7 | 6
  Phosphate; Grade 2 | 15 | 42
  Phosphate; Grade 3 | 5 | 8
  Phosphate; Grade 4 | 0 | 0
  Potassium; Grade 1 | 16 | 20
  Potassium; Grade 2 | 1 | 1
  Potassium; Grade 3 | 2 | 3
  Potassium; Grade 4 | 1 | 1
  Sodium; Grade 1 | 76 | 117
  Sodium; Grade 2 | 5 | 2
  Sodium; Grade 3 | 1 | 0
  Sodium; Grade 4 | 1 | 0
  Cholesterol; Grade 1 | 14 | 46
  Cholesterol; Grade 2 | 5 | 32
  Cholesterol; Grade 3 | 3 | 4
  Cholesterol; Grade 4 | 0 | 0
  Creatinine; Grade 1 | 1 | 4
  Creatinine; Grade 2 | 2 | 5
  Creatinine; Grade 3 | 0 | 0
  Creatinine; Grade 4 | 0 | 0
  Serum Triglycerides; Grade 1 | 0 | 0
  Serum Triglycerides; Grade 2 | 1 | 11
  Serum Triglycerides; Grade 3 | 1 | 3
  Serum Triglycerides; Grade 4 | 1 | 2

21. Secondary Outcome: Number of Participants With Clinical Chemistry Toxicities-Continuation Phase
Description: as for outcome 20
Time Frame: Up to Week 295
Population: Safety Continuation Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG in Continuation Phase
Number analyzed (Participants) | 274
Participants
  Serum glucose; Grade 1 | 43
  Serum glucose; Grade 2 | 33
  Serum glucose; Grade 3 | 9
  Serum glucose; Grade 4 | 0
  ALT; Grade 1 | 46
  ALT; Grade 2 | 16
  ALT; Grade 3 | 2
  ALT; Grade 4 | 0
  Albumin; Grade 1 | 1
  Albumin; Grade 2 | 4
  Albumin; Grade 3 | 0
  Albumin; Grade 4 | 0
  ALP; Grade 1 | 13
  ALP; Grade 2 | 2
  ALP; Grade 3 | 0
  ALP; Grade 4 | 0
  AST; Grade 1 | 37
  AST; Grade 2 | 11
  AST; Grade 3 | 5
  AST; Grade 4 | 1
  Bilirubin; Grade 1 | 14
  Bilirubin; Grade 2 | 9
  Bilirubin; Grade 3 | 0
  Bilirubin; Grade 4 | 2
  CO2; Grade 1 | 83
  CO2; Grade 2 | 20
  CO2; Grade 3 | 0
  CO2; Grade 4 | 0
  Creatine kinase; Grade 1 | 24
  Creatine kinase; Grade 2 | 6
  Creatine kinase; Grade 3 | 5
  Creatine kinase; Grade 4 | 5
  LDL cholesterol calculation; Grade 1 | 1
  LDL cholesterol calculation; Grade 2 | 1
  LDL cholesterol calculation; Grade 3 | 0
  LDL cholesterol calculation; Grade 4 | 0
  LDL cholesterol direct; Grade 1 | 1
  LDL cholesterol direct; Grade 2 | 1
  LDL cholesterol direct; Grade 3 | 0
  LDL cholesterol direct; Grade 4 | 0
  Lipase; Grade 1 | 19
  Lipase; Grade 2 | 9
  Lipase; Grade 3 | 2
  Lipase; Grade 4 | 4
  Phosphate; Grade 1 | 16
  Phosphate; Grade 2 | 38
  Phosphate; Grade 3 | 6
  Phosphate; Grade 4 | 0
  Potassium; Grade 1 | 24
  Potassium; Grade 2 | 5
  Potassium; Grade 3 | 1
  Potassium; Grade 4 | 1
  Sodium; Grade 1 | 69
  Sodium; Grade 2 | 0
  Sodium; Grade 3 | 0
  Sodium; Grade 4 | 0
  Cholesterol; Grade 1 | 1
  Cholesterol; Grade 2 | 0
  Cholesterol; Grade 3 | 1
  Cholesterol; Grade 4 | 0
  Creatinine; Grade 1 | 7
  Creatinine; Grade 2 | 4
  Creatinine; Grade 3 | 0
  Creatinine; Grade 4 | 0
  Serum Triglycerides; Grade 1 | 0
  Serum Triglycerides; Grade 2 | 0
  Serum Triglycerides; Grade 3 | 0
  Serum Triglycerides; Grade 4 | 1

22. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes. Change from Baseline in clinical hematology parameters at Weeks 4, 8, 16, 24, 36, 48, 52 are presented. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 8, Week 16, Week 24, Week 36, Week 48 and Week 52
Population: Safety Population. Two participants who were randomized to receive LPV/RTV received DTG and were included in DTG group for Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
10^9 cells/liter
  Basophil; Week 4; n= 289, 291: number analyzed (Participants) | 289 | 291
  Basophil; Week 4; n= 289, 291 | 0.00 (0.029) | 0.00 (0.016)
  Basophil; Week 8; n= 296, 289: number analyzed (Participants) | 296 | 289
  Basophil; Week 8; n= 296, 289 | 0.00 (0.017) | 0.00 (0.017)
  Basophil; Week 16; n= 286, 286: number analyzed (Participants) | 286 | 286
  Basophil; Week 16; n= 286, 286 | 0.00 (0.017) | 0.00 (0.017)
  Basophil; Week 24; n= 290, 281: number analyzed (Participants) | 290 | 281
  Basophil; Week 24; n= 290, 281 | 0.01 (0.017) | 0.00 (0.017)
  Basophil; Week 36; n= 283, 275: number analyzed (Participants) | 283 | 275
  Basophil; Week 36; n= 283, 275 | 0.01 (0.021) | 0.00 (0.018)
  Basophil; Week 48; n= 266, 242: number analyzed (Participants) | 266 | 242
  Basophil; Week 48; n= 266, 242 | 0.01 (0.021) | 0.01 (0.019)
  Basophil; Week 52; n= 265, 229: number analyzed (Participants) | 265 | 229
  Basophil; Week 52; n= 265, 229 | 0.01 (0.018) | 0.01 (0.022)
  Eosinophil; Week 4; n= 290, 291: number analyzed (Participants) | 290 | 291
  Eosinophil; Week 4; n= 290, 291 | 0.02 (0.182) | 0.02 (0.287)
  Eosinophil; Week 8; n= 296, 289: number analyzed (Participants) | 296 | 289
  Eosinophil; Week 8; n= 296, 289 | 0.03 (0.281) | 0.01 (0.175)
  Eosinophil; Week 16; n= 286, 286: number analyzed (Participants) | 286 | 286
  Eosinophil; Week 16; n= 286, 286 | 0.01 (0.240) | 0.01 (0.201)
  Eosinophil; Week 24; n= 290, 281: number analyzed (Participants) | 290 | 281
  Eosinophil; Week 24; n= 290, 281 | 0.02 (0.188) | 0.01 (0.173)
  Eosinophil; Week 36; n= 283, 275: number analyzed (Participants) | 283 | 275
  Eosinophil; Week 36; n= 283, 275 | 0.04 (0.214) | 0.02 (0.192)
  Eosinophil; Week 48; n= 266, 242: number analyzed (Participants) | 266 | 242
  Eosinophil; Week 48; n= 266, 242 | 0.04 (0.267) | 0.01 (0.210)
  Eosinophil; Week 52; n= 265, 229: number analyzed (Participants) | 265 | 229
  Eosinophil; Week 52; n= 265, 229 | 0.02 (0.188) | 0.01 (0.217)
  Lymphocyte; Week 4; n= 289, 291: number analyzed (Participants) | 289 | 291
  Lymphocyte; Week 4; n= 289, 291 | 0.13 (0.519) | 0.10 (0.549)
  Lymphocyte; Week 8; n= 296, 289: number analyzed (Participants) | 296 | 289
  Lymphocyte; Week 8; n= 296, 289 | 0.23 (0.592) | 0.29 (0.651)
  Lymphocyte; Week 16; n= 286, 286: number analyzed (Participants) | 286 | 286
  Lymphocyte; Week 16; n= 286, 286 | 0.28 (0.611) | 0.29 (0.668)
  Lymphocyte; Week 24; n= 290, 281: number analyzed (Participants) | 290 | 281
  Lymphocyte; Week 24; n= 290, 281 | 0.31 (0.589) | 0.34 (0.625)
  Lymphocyte; Week 36; n= 283, 275: number analyzed (Participants) | 283 | 275
  Lymphocyte; Week 36; n= 283, 275 | 0.38 (0.595) | 0.35 (0.646)
  Lymphocyte; Week 48; n= 266, 242: number analyzed (Participants) | 266 | 242
  Lymphocyte; Week 48; n= 266, 242 | 0.38 (0.648) | 0.37 (0.697)
  Lymphocyte; Week 52; n= 265, 229: number analyzed (Participants) | 265 | 229
  Lymphocyte; Week 52; n= 265, 229 | 0.34 (0.716) | 0.39 (0.720)
  Monocyte; Week 4; n= 289, 291: number analyzed (Participants) | 289 | 291
  Monocyte; Week 4; n= 289, 291 | 0.02 (0.201) | 0.00 (0.167)
  Monocyte; Week 8; n= 296, 289: number analyzed (Participants) | 296 | 289
  Monocyte; Week 8; n= 296, 289 | 0.01 (0.159) | 0.02 (0.174)
  Monocyte; Week 16; n= 286, 286: number analyzed (Participants) | 286 | 286
  Monocyte; Week 16; n= 286, 286 | -0.00 (0.140) | 0.01 (0.154)
  Monocyte; Week 24; n= 290, 281: number analyzed (Participants) | 290 | 281
  Monocyte; Week 24; n= 290, 281 | -0.01 (0.139) | 0.01 (0.173)
  Monocyte; Week 36; n= 283, 275: number analyzed (Participants) | 283 | 275
  Monocyte; Week 36; n= 283, 275 | 0.01 (0.151) | 0.02 (0.175)
  Monocyte; Week 48; n= 266, 242: number analyzed (Participants) | 266 | 242
  Monocyte; Week 48; n= 266, 242 | 0.01 (0.157) | 0.03 (0.190)
  Monocyte; Week 52; n= 265, 229: number analyzed (Participants) | 265 | 229
  Monocyte; Week 52; n= 265, 229 | 0.01 (0.173) | 0.02 (0.205)
  Neutrophil; Week 4; n= 289, 291: number analyzed (Participants) | 289 | 291
  Neutrophil; Week 4; n= 289, 291 | 0.35 (1.914) | 0.23 (1.407)
  Neutrophil; Week 8; n= 296, 289: number analyzed (Participants) | 296 | 289
  Neutrophil; Week 8; n= 296, 289 | 0.27 (1.491) | 0.23 (1.678)
  Neutrophil; Week 16; n= 286, 286: number analyzed (Participants) | 286 | 286
  Neutrophil; Week 16; n= 286, 286 | 0.31 (1.462) | 0.29 (1.481)
  Neutrophil; Week 24; n= 290, 281: number analyzed (Participants) | 290 | 281
  Neutrophil; Week 24; n= 290, 281 | 0.42 (1.694) | 0.34 (1.315)
  Neutrophil; Week 36; n= 283, 275: number analyzed (Participants) | 283 | 275
  Neutrophil; Week 36; n= 283, 275 | 0.50 (1.605) | 0.37 (1.661)
  Neutrophil; Week 48; n= 266, 242: number analyzed (Participants) | 266 | 242
  Neutrophil; Week 48; n= 266, 242 | 0.46 (1.491) | 0.50 (1.449)
  Neutrophil; Week 52; n= 265, 229: number analyzed (Participants) | 265 | 229
  Neutrophil; Week 52; n= 265, 229 | 0.63 (1.691) | 0.44 (1.604)
  Platelet; Week 4; n= 291, 293: number analyzed (Participants) | 291 | 293
  Platelet; Week 4; n= 291, 293 | 22.81 (63.368) | 23.64 (53.514)
  Platelet; Week 8; n= 293, 293: number analyzed (Participants) | 293 | 293
  Platelet; Week 8; n= 293, 293 | 22.95 (62.969) | 26.17 (58.634)
  Platelet; Week 16; n= 287, 286: number analyzed (Participants) | 287 | 286
  Platelet; Week 16; n= 287, 286 | 21.77 (66.974) | 28.03 (61.780)
  Platelet; Week 24; n= 290, 282: number analyzed (Participants) | 290 | 282
  Platelet; Week 24; n= 290, 282 | 19.79 (63.702) | 27.32 (65.103)
  Platelet; Week 36; n= 283, 274: number analyzed (Participants) | 283 | 274
  Platelet; Week 36; n= 283, 274 | 20.02 (69.570) | 21.41 (64.787)
  Platelet; Week 48; n= 265, 246: number analyzed (Participants) | 265 | 246
  Platelet; Week 48; n= 265, 246 | 16.72 (66.983) | 30.20 (63.038)
  Platelet; Week 52; n= 267, 232: number analyzed (Participants) | 267 | 232
  Platelet; Week 52; n= 267, 232 | 20.98 (66.402) | 32.60 (71.882)
  Leukocyte; Week 4; n= 289, 292: number analyzed (Participants) | 289 | 292
  Leukocyte; Week 4; n= 289, 292 | 0.51 (2.105) | 0.37 (1.607)
  Leukocyte; Week 8; n= 296, 292: number analyzed (Participants) | 296 | 292
  Leukocyte; Week 8; n= 296, 292 | 0.54 (1.676) | 0.54 (1.879)
  Leukocyte; Week 16; n= 290, 288: number analyzed (Participants) | 290 | 288
  Leukocyte; Week 16; n= 290, 288 | 0.61 (1.622) | 0.60 (1.746)
  Leukocyte; Week 24; n= 291, 284: number analyzed (Participants) | 291 | 284
  Leukocyte; Week 24; n= 291, 284 | 0.75 (1.826) | 0.70 (1.545)
  Leukocyte; Week 36; n= 285, 276: number analyzed (Participants) | 285 | 276
  Leukocyte; Week 36; n= 285, 276 | 0.91 (1.777) | 0.76 (1.913)
  Leukocyte; Week 48; n= 267, 245: number analyzed (Participants) | 267 | 245
  Leukocyte; Week 48; n= 267, 245 | 0.91 (1.777) | 0.90 (1.718)
  Leukocyte; Week 52; 268, 231: number analyzed (Participants) | 268 | 231
  Leukocyte; Week 52; 268, 231 | 0.99 (1.908) | 0.86 (1.819)

23. Secondary Outcome: Change From Baseline in Hematocrit Values
Description: Blood samples were collected from participants to evaluate clinical hematology parameter including hematocrit. Change from Baseline in hematocrit values at Weeks 4, 8, 16, 24, 36, 48, 52 are presented. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 8, Week 16, Week 24, Week 36, Week 48 and and Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Proportion of red blood cells in blood
  Week 4; n= 296, 296: number analyzed (Participants) | 296 | 296
  Week 4; n= 296, 296 | -0.00 (0.032) | -0.01 (0.029)
  Week 8; n= 297, 294: number analyzed (Participants) | 297 | 294
  Week 8; n= 297, 294 | 0.00 (0.039) | -0.01 (0.037)
  Week 16; n= 290, 289: number analyzed (Participants) | 290 | 289
  Week 16; n= 290, 289 | 0.01 (0.044) | -0.01 (0.042)
  Week 24; n= 291, 285: number analyzed (Participants) | 291 | 285
  Week 24; n= 291, 285 | 0.01 (0.037) | -0.00 (0.039)
  Week 36; n= 286, 276: number analyzed (Participants) | 286 | 276
  Week 36; n= 286, 276 | 0.01 (0.038) | -0.00 (0.039)
  Week 48; n= 268, 248: number analyzed (Participants) | 268 | 248
  Week 48; n= 268, 248 | 0.02 (0.038) | -0.00 (0.041)
  Week 52; n= 269, 233: number analyzed (Participants) | 269 | 233
  Week 52; n= 269, 233 | 0.02 (0.040) | -0.00 (0.041)

24. Secondary Outcome: Change From Baseline in Hemoglobin Values
Description: Blood samples were collected from participants to evaluate clinical hematology parameter including hemoglobin. Change from Baseline in hemoglobin values at Weeks 4, 8, 16, 24, 36, 48, 52 are presented. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 8, Week 16, Week 24, Week 36, Week 48 and Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Gram per liter
  Week 4; n= 296, 296: number analyzed (Participants) | 296 | 296
  Week 4; n= 296, 296 | -1.33 (9.858) | -4.23 (8.994)
  Week 8; n= 297, 294: number analyzed (Participants) | 297 | 294
  Week 8; n= 297, 294 | -0.12 (11.725) | -4.41 (11.340)
  Week 16; n= 290, 289: number analyzed (Participants) | 290 | 289
  Week 16; n= 290, 289 | 2.39 (12.905) | -2.10 (12.904)
  Week 24; n= 291, 285: number analyzed (Participants) | 291 | 285
  Week 24; n= 291, 285 | 3.05 (10.881) | -0.46 (12.363)
  Week 36; n= 286, 276: number analyzed (Participants) | 286 | 276
  Week 36; n= 286, 276 | 5.18 (11.968) | 0.34 (12.628)
  Week 48; n= 268, 248: number analyzed (Participants) | 268 | 248
  Week 48; n= 268, 248 | 6.05 (12.138) | 0.90 (13.486)
  Week 52; n= 269, 233: number analyzed (Participants) | 269 | 233
  Week 52; n= 269, 233 | 5.68 (12.457) | 1.07 (13.361)

25. Secondary Outcome: Change From Baseline in Mean Corpuscular Volume (MCV)
Description: Blood samples were collected from participants to evaluate clinical hematology parameter including MCV. Change from Baseline in MCV values at Weeks 4, 8, 16, 24, 36, 48, 52 are presented. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 8, Week 16, Week 24, Week 36, Week 48 and and Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Femtoliter
  Week 4; n= 296, 296: number analyzed (Participants) | 296 | 296
  Week 4; n= 296, 296 | 0.68 (3.820) | 0.46 (3.799)
  Week 8; n= 297, 294: number analyzed (Participants) | 297 | 294
  Week 8; n= 297, 294 | 1.72 (7.659) | 1.78 (7.266)
  Week 16; n= 290, 289: number analyzed (Participants) | 290 | 289
  Week 16; n= 290, 289 | 3.91 (13.827) | 3.83 (13.600)
  Week 24; n= 291, 285: number analyzed (Participants) | 291 | 285
  Week 24; n= 291, 285 | 4.86 (15.279) | 4.39 (15.099)
  Week 36; n= 286, 276: number analyzed (Participants) | 286 | 276
  Week 36; n= 286, 276 | 4.33 (15.450) | 4.62 (15.413)
  Week 48; n= 268, 248: number analyzed (Participants) | 268 | 248
  Week 48; n= 268, 248 | 4.14 (15.637) | 4.79 (15.463)
  Week 52; n= 269, 233: number analyzed (Participants) | 269 | 233
  Week 52; n= 269, 233 | 4.36 (15.496) | 4.72 (15.697)

26. Secondary Outcome: Change From Baseline in Erythrocyte Values
Description: Blood samples were collected from participants to evaluate clinical hematology parameter including erythrocyte. Change from Baseline in erythrocyte values at Weeks 4, 8, 16, 24, 36, 48, 52 are presented. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 8, Week 16, Week 24, Week 36, Week 48 and up to Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
10^12 cells/liter
  Week 4; n= 296, 296: number analyzed (Participants) | 296 | 296
  Week 4; n= 296, 296 | -0.08 (0.385) | -0.16 (0.363)
  Week 8; n= 297, 294: number analyzed (Participants) | 297 | 294
  Week 8; n= 297, 294 | -0.07 (0.558) | -0.23 (0.529)
  Week 16; n= 290, 289: number analyzed (Participants) | 290 | 289
  Week 16; n= 290, 289 | -0.06 (0.808) | -0.21 (0.754)
  Week 24; n= 291, 285: number analyzed (Participants) | 291 | 285
  Week 24; n= 291, 285 | -0.08 (0.768) | -0.20 (0.747)
  Week 36; n= 286, 276: number analyzed (Participants) | 286 | 276
  Week 36; n= 286, 276 | -0.01 (0.792) | -0.18 (0.749)
  Week 48; n= 268, 248: number analyzed (Participants) | 268 | 248
  Week 48; n= 268, 248 | 0.01 (0.798) | -0.18 (0.750)
  Week 52; n= 269, 233: number analyzed (Participants) | 269 | 233
  Week 52; n= 269, 233 | -0.01 (0.788) | -0.17 (0.761)

27. Secondary Outcome: Number of Participants With Hematology Toxicities -Randomized Phase
Description: Number of participants with hematology toxicities has been presented. Toxicities were based on the Division of AIDS (DAIDS) grading system. Grade 1=Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Potentially life-threatening. Higher the grade, more severe the symptoms. Data has been reported for hematology parameters including Hemoglobin, Leukocytes, Neutrophils and Platelets.
Time Frame: Up to Week 52
Population: Safety Population. Two participants who were randomized to receive LPV/RTV received DTG and were included in DTG group for Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Participants
  Hemoglobin; Grade 1 | 6 | 18
  Hemoglobin; Grade 2 | 5 | 4
  Hemoglobin; Grade 3 | 5 | 0
  Hemoglobin; Grade 4 | 4 | 1
  Leukocytes; Grade 1 | 19 | 10
  Leukocytes; Grade 2 | 5 | 5
  Leukocytes; Grade 3 | 3 | 0
  Leukocytes; Grade 4 | 0 | 0
  Neutrophils; Grade 1 | 25 | 26
  Neutrophils; Grade 2 | 9 | 11
  Neutrophils; Grade 3 | 10 | 3
  Neutrophils; Grade 4 | 4 | 0
  Platelets; Grade 1 | 6 | 4
  Platelets; Grade 2 | 2 | 7
  Platelets; Grade 3 | 0 | 1
  Platelets; Grade 4 | 1 | 0

28. Secondary Outcome: Number of Participants With Hematology Toxicities-Continuation Phase
Description: as for outcome 27
Time Frame: Up to Week 295
Population: Safety-Continuation Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG in Continuation Phase
Number analyzed (Participants) | 274
Participants
  Hemoglobin; Grade 1 | 13
  Hemoglobin; Grade 2 | 2
  Hemoglobin; Grade 3 | 1
  Hemoglobin; Grade 4 | 0
  Leukocytes; Grade 1 | 23
  Leukocytes; Grade 2 | 6
  Leukocytes; Grade 3 | 0
  Leukocytes; Grade 4 | 0
  Neutrophils; Grade 1 | 21
  Neutrophils; Grade 2 | 16
  Neutrophils; Grade 3 | 10
  Neutrophils; Grade 4 | 2
  Platelets; Grade 1 | 6
  Platelets; Grade 2 | 3
  Platelets; Grade 3 | 1
  Platelets; Grade 4 | 0

29. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to AEs-Randomized Phase
Description: Number of participants who discontinued study treatment due to AEs or SAEs were summarized.
Time Frame: Up to Week 52
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Participants | 8 | 18

30. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to AEs-Continuation Phase
Description: Number of participants who discontinued study treatment due to AEs were summarized.
Time Frame: Up to Week 295
Population: Safety-Continuation Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG in Continuation Phase
Number analyzed (Participants) | 274
Participants | 9

31. Secondary Outcome: Change From Baseline in Fasting LDL Cholesterol at Week 24 and Week 48
Description: Blood samples were collected from participants in fasting state to evaluate LDL cholesterol. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value. Analysis was performed using multiple imputation with missing at random assumption. Only participants available at the time of evaluation were analyzed.
Time Frame: Baseline (Day 1, Pre-dose), Week 24 and Week 48
Population: Safety Population. Only those participants with data available at specified time points were analyzed. Two participants who were randomized to receive LPV/RTV received DTG and were included in DTG group for Safety Population.
Measure: Mean (Standard Error); unit: Millimoles per liter
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 303 | 292
Millimoles per liter
  Week 24 | -0.121 (0.0356) | 0.050 (0.0378)
  Week 48 | -0.012 (0.0387) | 0.135 (0.0416)
Statistical Analysis 1: Comparison: Participants Receiving DTG-Randomized Phase vs Participants Receiving LPV/RTV-Randomized Phase; Test type: Other; p = 0.0010, Multiple imputation; Mean Difference (Net) = -0.171, 95% CI 2-sided [-0.272 to -0.069] — Mean difference at Week 24 was calculated using multiple imputation using missing at random, adjusting for Baseline LDL cholesterol, Baseline plasma HIV-1 RNA, Baseline number of Fully Active NRTIs in the background regimen and Age
Statistical Analysis 2: Comparison: Participants Receiving DTG-Randomized Phase vs Participants Receiving LPV/RTV-Randomized Phase; Test type: Other; p = 0.0100, 'Multiple imputation; Mean Difference (Net) = -0.147, 95% CI 2-sided [-0.259 to -0.035] — Mean difference at Week 48 was calculated using multiple imputation using missing at random, adjusting for Baseline LDL cholesterol, Baseline plasma HIV-1 RNA, Baseline number of Fully Active NRTIs in the background regimen and Age

32. Secondary Outcome: Change From Baseline in Fasting Total Cholesterol/HDL Cholesterol Ratio
Description: Blood samples were collected from participants in fasting state to evaluate total cholesterol/HDL cholesterol ratio. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value. Only participants available at the time of evaluation were analyzed. Analysis was performed using multiple imputation with missing at random assumption.
Time Frame: Baseline (Day 1, Pre-dose), Week 24 and Week 48
Population: Safety Population. Only those participants with data available at specified time point were analyzed. Two participants who were randomized to receive LPV/RTV received DTG and were included in DTG group for Safety Population.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 306 | 295
Ratio
  Week 24 | -0.237 (0.0662) | 0.305 (0.0683)
  Week 48 | -0.084 (0.0693) | 0.275 (0.0729)
Statistical Analysis 1: Comparison: Participants Receiving DTG-Randomized Phase vs Participants Receiving LPV/RTV-Randomized Phase; Test type: Other; p < 0.0001, Multiple imputation; Mean Difference (Net) = -0.542, 95% CI 2-sided [-0.729 to -0.356] — Estimates at Week 24 are calculated using multiple imputation using missing at random, adjusting for Baseline total cholesterol/HDL ratio, Baseline plasma HIV-1 RNA, Baseline number of Fully Active NRTIs in the background regimen and Age
Statistical Analysis 2: Comparison: Participants Receiving DTG-Randomized Phase vs Participants Receiving LPV/RTV-Randomized Phase; Test type: Other; p = 0.0004, Multiple imputation; Mean Difference (Net) = -0.358, 95% CI 2-sided [-0.555 to -0.161] — Estimates at Week 48 are calculated using multiple imputation using missing at random, adjusting for Baseline total cholesterol/HDL ratio, Baseline plasma HIV-1 RNA, Baseline number of Fully Active NRTIs in the background regimen and Age

33. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Grade 2 or Greater Laboratory Abnormalities in Fasting LDL Cholesterol
Description: Blood samples were collected from participants in fasting state at indicated time-points to evaluate LDL cholesterol. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value. Number of participants who experienced maximum grade 2 or greater toxicity post-Baseline in fasting LDL cholesterol was summarized. Participants were graded using the Division of AIDS Table for Grading Severity of Adult and Pediatric Adverse Events. Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=potentially life-threatening. Higher the grade, more severe the symptoms.
Time Frame: Up to Week 48
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Participants | 5 | 20

34. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Grade 2 or Greater Drug-related Diarrhea
Description: Number of participants who experienced maximum grade 2 or greater toxicity post-Baseline in drug-related diarrhea was summarized. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value. Participants were graded using the Division of AIDS Table for Grading Severity of Adult and Pediatric Adverse Events. Grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=potentially life-threatening. Higher the grade, more severe the symptoms.
Time Frame: Week 24 and Week 48
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 314 | 310
Participants
  Week 24 | 1 | 22
  Week 48 | 1 | 23

35. Secondary Outcome: Change From Baseline in Gastrointestinal Symptom Rating Scale (GSRS) Score
Description: The GSRS is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhea and Constipation. The scale ranges from 1= no discomfort to 7= very severe discomfort for each symptom cluster. Higher scores show greater severity of symptoms. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value. The analysis was performed using Last Observation Carried Forward (LOCF) dataset. In the LOCF dataset, missing values were carried forward from the previous, non-missing available on-treatment assessment.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 24, Week 48
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 312 | 312
Scores on a scale
  Diarrhea Syndrome Score; Week 4; n= 303, 305: number analyzed (Participants) | 303 | 305
  Diarrhea Syndrome Score; Week 4; n= 303, 305 | 0.00 [-0.33 to 0.00] | 0.00 [0.00 to 1.33]
  Diarrhea Syndrome Score; Week 24; n= 305, 306: number analyzed (Participants) | 305 | 306
  Diarrhea Syndrome Score; Week 24; n= 305, 306 | 0.00 [-0.33 to 0.00] | 0.00 [0.00 to 1.00]
  Diarrhea Syndrome Score; Week 48; n= 305, 306: number analyzed (Participants) | 305 | 306
  Diarrhea Syndrome Score; Week 48; n= 305, 306 | 0.00 [-0.33 to 0.00] | 0.00 [0.00 to 0.67]
  Indigestion Syndrome Score; Week 4; n=305, 306: number analyzed (Participants) | 305 | 306
  Indigestion Syndrome Score; Week 4; n=305, 306 | 0.00 [-0.25 to 0.00] | 0.00 [0.00 to 0.75]
  Indigestion Syndrome Score; Week 24; n= 306, 307: number analyzed (Participants) | 306 | 307
  Indigestion Syndrome Score; Week 24; n= 306, 307 | 0.00 [-0.25 to 0.00] | 0.00 [-0.25 to 0.50]
  Indigestion Syndrome Score; Week 48; n= 306, 307: number analyzed (Participants) | 306 | 307
  Indigestion Syndrome Score; Week 48; n= 306, 307 | 0.00 [-0.50 to 0.00] | 0.00 [-0.25 to 0.50]
  Constipation Score; Week 4; n= 305, 305: number analyzed (Participants) | 305 | 305
  Constipation Score; Week 4; n= 305, 305 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.33]
  Constipation Score; Week 24; n= 306, 306: number analyzed (Participants) | 306 | 306
  Constipation Score; Week 24; n= 306, 306 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.33]
  Constipation Score; Week 48; n= 306, 306: number analyzed (Participants) | 306 | 306
  Constipation Score; Week 48; n= 306, 306 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.33]
  Abdominal pain Score; Week 4; n= 305, 306: number analyzed (Participants) | 305 | 306
  Abdominal pain Score; Week 4; n= 305, 306 | 0.00 [-0.33 to 0.00] | 0.00 [0.00 to 0.67]
  Abdominal pain Score; Week 24; n= 306, 307: number analyzed (Participants) | 306 | 307
  Abdominal pain Score; Week 24; n= 306, 307 | 0.00 [-0.33 to 0.00] | 0.00 [-0.33 to 0.67]
  Abdominal pain Score; Week 48; n= 306, 307: number analyzed (Participants) | 306 | 307
  Abdominal pain Score; Week 48; n= 306, 307 | 0.00 [-0.67 to 0.00] | 0.00 [0.00 to 0.33]
  Reflux Score; Week 4; n= 305, 306: number analyzed (Participants) | 305 | 306
  Reflux Score; Week 4; n= 305, 306 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.50]
  Reflux Score; Week 24; n= 306, 307: number analyzed (Participants) | 306 | 307
  Reflux Score; Week 24; n= 306, 307 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Reflux Score; Week 48; n= 306, 307: number analyzed (Participants) | 306 | 307
  Reflux Score; Week 48; n= 306, 307 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.50]

36. Secondary Outcome: Change From Baseline in Treatment Satisfaction, Using the HIV-Treatment Satisfaction Questionnaire (HIVTSQ) Score
Description: The HIVTSQ is a self-reported scales that measure overall satisfaction with treatment. The score ranges from 0-10. The higher the score, the greater the improvement in treatment satisfaction as compared to the past few weeks. A smaller score represents a decline in treatment satisfaction compared to the past few weeks. Baseline was defined as the latest pre-dose assessment value. Change from Baseline was calculated as post-Baseline visit values minus Baseline value. The analysis was performed using LOCF dataset. In the LOCF dataset, missing values were carried forward from the previous, non-missing available on-treatment assessment.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 24, Week 48
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 312 | 312
Scores on a scale
  Week 4; n= 304, 306: number analyzed (Participants) | 304 | 306
  Week 4; n= 304, 306 | 3.4 [0.0 to 11.5] | 2.0 [0.0 to 10.0]
  Week 24; n= 305, 307: number analyzed (Participants) | 305 | 307
  Week 24; n= 305, 307 | 5.0 [0.0 to 13.0] | 3.0 [0.0 to 12.0]
  Week 48; n= 305, 307: number analyzed (Participants) | 305 | 307
  Week 48; n= 305, 307 | 5.0 [0.0 to 14.0] | 3.0 [0.0 to 11.0]

37. Secondary Outcome: Number of Participants Showing Adherence With Treatment, Using the Morisky 8-Item Medication Adherence Scale (MMAS-8)
Description: Treatment compliance was evaluated through MMAS-8. It is an eight-item self-reported measure of medication-taking behavior. The score ranges from 0-8 where scores of 8 indicate high or near perfect adherence, and scores of less than 6 indicate poor or inadequate adherence on the MMAS-8 scale. Number of participants showing low, medium and high adherence to treatment are presented. Low adherence is a score 0-5.75, medium adherence is a score of 6-7.75 and high adherence is a score of 8. The analysis was performed using LOCF dataset. In the LOCF dataset, missing values were carried forward from the previous, non-missing available on-treatment assessment.
Time Frame: Baseline (Day 1, Pre-dose), Week 4, Week 24 and Week 48
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase
Number analyzed (Participants) | 312 | 312
Participants
  Baseline (Day 1, Pre-dose); low; n= 309, 312: number analyzed (Participants) | 309 | 312
  Baseline (Day 1, Pre-dose); low; n= 309, 312 | 70 | 75
  Baseline (Day 1, Pre-dose); medium; n= 309, 312: number analyzed (Participants) | 309 | 312
  Baseline (Day 1, Pre-dose); medium; n= 309, 312 | 102 | 100
  Baseline (Day 1, Pre-dose); high; n= 309, 312: number analyzed (Participants) | 309 | 312
  Baseline (Day 1, Pre-dose); high; n= 309, 312 | 137 | 137
  Week 4; low; n= 306, 306: number analyzed (Participants) | 306 | 306
  Week 4; low; n= 306, 306 | 17 | 37
  Week 4; medium; n= 306, 306: number analyzed (Participants) | 306 | 306
  Week 4; medium; n= 306, 306 | 81 | 80
  Week 4; high n= 306, 306: number analyzed (Participants) | 306 | 306
  Week 4; high n= 306, 306 | 208 | 189
  Week 24; low; n= 307, 307: number analyzed (Participants) | 307 | 307
  Week 24; low; n= 307, 307 | 25 | 39
  Week 24; medium; n= 307, 307: number analyzed (Participants) | 307 | 307
  Week 24; medium; n= 307, 307 | 83 | 76
  Week 24; high; n= 307,307: number analyzed (Participants) | 307 | 307
  Week 24; high; n= 307,307 | 199 | 192
  Week 48; low; n= 307, 307: number analyzed (Participants) | 307 | 307
  Week 48; low; n= 307, 307 | 28 | 52
  Week 48; medium; n= 307, 307: number analyzed (Participants) | 307 | 307
  Week 48; medium; n= 307, 307 | 74 | 82
  Week 48; high; n= 307, 307: number analyzed (Participants) | 307 | 307
  Week 48; high; n= 307, 307 | 205 | 173

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious adverse events (SAEs) and non-SAEs were collected up to Week 52 for Randomized Phase; up to Week 295 for Continuation Phase and up to Week 348 for Randomized Phase+Continuation Phase.
Description: All-cause mortality, SAEs and non-SAEs were reported for the Safety Population for the Randomized Phase and Randomized + Continuation Phase. Two participants who were randomized to receive LPV/RTV received DTG and were included in DTG group for Safety Population. Safety-Continuation Population was used for the Continuation Phase.
Arm/Group | Participants Receiving DTG-Randomized Phase | Participants Receiving LPV/RTV-Randomized Phase | Participants Receiving DTG-Continuation Phase | DTG in Randomized Phase Followed by Continuation Phase | LPV/RTV-Randomized Phase Followed by DTG in Continuation Phase
All-Cause Mortality (participants affected / at risk) | 2/314 | 3/310 | 3/274 | 5/314 | 3/310
Serious Adverse Events (participants affected / at risk) | 20/314 | 20/310 | 29/274 | 47/314 | 20/310
Other Adverse Events (participants affected / at risk) | 155/314 | 202/310 | 150/274 | 218/314 | 213/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Receiving DTG-Randomized Phase (N=314) | Participants Receiving LPV/RTV-Randomized Phase (N=310) | Participants Receiving DTG-Continuation Phase (N=274) | DTG in Randomized Phase Followed by Continuation Phase (N=314) | LPV/RTV-Randomized Phase Followed by DTG in Continuation Phase (N=310)
Pneumonia (Infections and infestations) | 3 (3) | 5 (5) | 0 (0) | 3 (3) | 5 (5)
Cerebral toxoplasmosis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Bone tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus chorioretinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Extrapulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Immune reconstitution inflammatory syndrome associated tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Intestinal tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leptospirosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Secondary syphilis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tuberculosis gastrointestinal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Receiving DTG-Randomized Phase (N=314) | Participants Receiving LPV/RTV-Randomized Phase (N=310) | Participants Receiving DTG-Continuation Phase (N=274) | DTG in Randomized Phase Followed by Continuation Phase (N=314) | LPV/RTV-Randomized Phase Followed by DTG in Continuation Phase (N=310)
Diarrhoea (Gastrointestinal disorders) | 28 (35) | 105 (134) | 19 (25) | 38 (54) | 105 (134)
Nausea (Gastrointestinal disorders) | 10 (11) | 30 (33) | 5 (6) | 14 (16) | 30 (33)
Vomiting (Gastrointestinal disorders) | 5 (5) | 21 (24) | 2 (4) | 6 (8) | 21 (24)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 12 (13) | 9 (12) | 19 (22) | 12 (13)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 8 (9) | 7 (8) | 16 (17) | 8 (9)
Flatulence (Gastrointestinal disorders) | 6 (7) | 8 (8) | 0 (0) | 6 (7) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 45 (59) | 43 (52) | 65 (122) | 83 (178) | 43 (52)
Lower respiratory tract infection (Infections and infestations) | 13 (20) | 14 (17) | 16 (28) | 22 (48) | 14 (17)
Nasopharyngitis (Infections and infestations) | 8 (9) | 12 (13) | 10 (11) | 17 (19) | 12 (13)
Influenza (Infections and infestations) | 7 (8) | 9 (10) | 12 (14) | 18 (22) | 9 (10)
Herpes zoster (Infections and infestations) | 5 (5) | 8 (8) | 0 (0) | 7 (8) | 8 (8)
Syphilis (Infections and infestations) | 7 (7) | 5 (5) | 6 (6) | 12 (12) | 5 (5)
Urinary tract infection (Infections and infestations) | 9 (10) | 2 (2) | 12 (15) | 18 (25) | 2 (2)
Headache (Nervous system disorders) | 24 (24) | 16 (17) | 13 (15) | 37 (39) | 16 (17)
Dizziness (Nervous system disorders) | 9 (9) | 10 (10) | 0 (0) | 9 (11) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 11 (13) | 10 (13) | 6 (6) | 17 (19) | 10 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (7) | 0 (0) | 3 (3) | 8 (8)
Fatigue (General disorders) | 7 (7) | 5 (5) | 0 (0) | 8 (9) | 5 (5)
Pyrexia (General disorders) | 7 (7) | 5 (5) | 0 (0) | 11 (11) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 10 (10) | 16 (18) | 27 (34) | 10 (10)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 13 (14) | 0 (0) | 10 (10) | 13 (14)
Insomnia (Psychiatric disorders) | 8 (8) | 7 (7) | 7 (7) | 14 (15) | 7 (7)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 7 (7) | 0 (0) | 2 (2) | 7 (7)
Gastroenteritis (Infections and infestations) | 3 (3) | 7 (8) | 8 (11) | 10 (14) | 7 (8)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 7 (7) | 8 (9) | 14 (16) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (7) | 12 (14) | 20 (25) | 7 (7)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 7 (7) | 4 (6)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 8 (8) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 6 (6)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 5 (5)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 8 (8) | 9 (9) | 4 (5)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 7 (7) | 6 (6)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 7 (7) | 4 (4)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 7 (7) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (14) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 19 (20) | 24 (27) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 7 (8) | 12 (14) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 10 (14) | 11 (15) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 5 (5) | 7 (8) | 6 (6)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 10 (13) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 10 (14) | 15 (19) | 6 (6)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT02227238/Prot_002.pdf
  • Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/38/NCT02227238/SAP_003.pdf